CLINICAL TRIAL: NCT03529578
Title: A Case Series to Investigate the Safety and Efficacy of Weekly Application of Dehydrated Human Amnion/Chorion Membrane in the Treatment of Pressure Ulcers
Brief Title: A Single Center, Prospective, Case Series of the Treatment of Pressure Ulcers and Decubitus Ulcers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MiMedx Group, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EFPU002
Record Dates: First submitted 2018-03-20; First posted 2018-05-18 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Pressure Ulcer
Keywords: Pressure Ulcer, Decubitus Ulcer
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dHACM (Experimental): Standard of Care plus Weekly Application of dHACM
  Interventions: Procedure: dHACM

INTERVENTIONS:
Procedure: dHACM — Dehydrated human amnion/chorion membrane (dHACM) product and is regulated as a Human Cells, Tissues and Cellular and Tissue Based Product (HCT/P) under Section 361 of the Public Health Service Act by the Food and Drug Administration (FDA)

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of dehydrated amnion/chorion membrane (dHACM) in the treatment of patients with stage II or III pressure ulcer and decubitus ulcers

ELIGIBILITY:
Inclusion Criteria:

1. Index ulcer characteristics:

   1. Index ulcer area after debridement is ≥ 2 cm² and ≤ 25 cm² at the randomization visit
   2. Ulcer must be Stage II or III as determined by the National Pressure Ulcer Advisory Panel (NPUAP) pressure ulcer staging system
2. Subject criteria must include:

   1. Age 18 or older
   2. The subject or their legally authorized representative provides consent and is willing and able to participate in all procedures and follow-up evaluations necessary to complete the study

Exclusion Criteria:

1. Index ulcer characteristics that will make subject ineligible for enrollment:

   1. Stage I or IV ulcers as determined by NPUAP pressure ulcer staging system
   2. Signs and symptoms of local infection
   3. Previous surgical procedure performed at site
   4. Known or suspected local skin malignancy at index ulcer site
   5. Prior radiation therapy treatment at the index ulcer site
2. Subject criteria that will make subject ineligible for enrollment:

   1. Presence of other diseases which, in the Opinion of the Investigator, may result in allograft failure or has experienced graft failure in the past (examples include: immune system disorders including Systemic Lupus Erythematosus (SLE), Fibromyalgia, Acquired Immunodeficiency Syndrome (AIDS) or HIV)
   2. Currently taking medications which in the opinion of the investigator may affect graft incorporation
   3. Allergy or known sensitivity to Aminoglycosides such as gentamicin sulfate and/or streptomycin sulfate
   4. Any condition(s) that in the opinion of the investigator may seriously compromises the subject's ability to participate in this study. Examples include: known history of poor adherence with medical treatment, current drug or alcohol abuse or a medical/psychiatric condition
   5. Pregnancy at enrollment or within last 6 months, women who are breastfeeding, or women of childbearing potential who are planning to become pregnant during the time of the study OR are unwilling/unable to use acceptable methods of contraception (birth control pills, barriers, or abstinence)
   6. Subjects currently enrolled in this study (i.e. concurrent enrollment in the study is prohibited)
   7. Subject has used any investigational drug(s) or therapeutic device(s) within 30 days preceding screening.
   8. Any pathology that would limit the blood supply and compromise healing
   9. Subject is a prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with complete wound closure of study ulcer | 8 Weeks
  The percentage of subjects with complete wound closure of the study ulcer

SECONDARY OUTCOMES:
Wound healing kinetics: Complete wound healing | 8 weeks
  Total time for complete wound healing
Wound healing kinetics: Weekly percentage of wounds with total closure | 8 weeks
  Percentage of wounds with total closure at each weekly visit time point
Wound healing kinetics: rate of closure/week | 8 weeks
  Rate of wound closure/week
Incidence of Treatment-Emergent Adverse Events [Safety] | 8 weeks
  The endpoints for safety will be reported as the frequencies of occurrence of each adverse event, the rate of adverse events per patient/month and time to each event; Both serious and non-serious adverse events will be recorded
Wound Infection Rate [Safety] | 8 weeks
  Additionally, wound infection rates will be noted throughout the course of the study

OTHER OUTCOMES:
Comparison of Quality of Life for subjects [Exploratory] | 8 weeks
  Comparison of Quality of Life for subjects after treatment; This data will be measured by the SF-12 Health Survey at three time points throughout the study (8 weeks): prior to treatment, at 4 weeks, and at the end of the trial.

CONTACTS AND LOCATIONS:
Overall Officials: David Mason, MD, Study Director — Chief Medical Officer
Locations (1):
- Infectious Disease Specialists of Atlanta, PC, Decatur, Georgia, United States